CLINICAL TRIAL: NCT00010725
Title: Effects of Herbal Antioxidants on Cardiovascular Disease in Older Blacks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000082-01P3 (NIH); P50AT000082-01 (NIH); P50AT000082-02 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Cardiovascular Diseases
Keywords: CVD
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MAK
Drug: Vitamin Supplements

SUMMARY:
The purpose of this study is to compare an herbal supplement, nonfood-derived vitamins, and placebo for the care of cardiovascular disease in high risk older African Americans.

DETAILED DESCRIPTION:
Older African Americans suffer from disproportionately high rates of cardiovascular disease (CVD) morbidity and mortality. In response to the health disparity between older African Americans and whites, national mandates have called for new research on innovative approaches to CVD prevention in this high risk population. Oxidative stress has recently been implicated in the pathogenesis of atherosclerotic CVD. Available evidence from epidemiological studies, clinical trials, and laboratory mechanistic studies indicate that antioxidant interventions may be useful in the prevention and treatment of atherosclerotic CVD in high risk older populations. Furthermore, it has been hypothesized that dietary or food sources of antioxidant nutrients may be more clinically effective than conventional nonfood-derived vitamin supplementation. Surveys indicate relatively high rates of complementary and alternative medicine (CAM) use, including herbal medicines, in older African Americans. Yet, with the exception of the previous clinical trials of the present Center team, there have been few controlled studies on CAM therapies in older African Americans and no previous controlled studies on efficacy and mechanisms of herbal antioxidants for the prevention of CVD in this high risk population. Preliminary studies have found that a CAM herbal preparation (MAK) derived from traditional Vedic medicine demonstrates potent antioxidant and anti-atherogenic effects in laboratory and pilot human studies. This study will evaluate the effects of this traditional CAM herbal preparation in older African Americans.

This will be a controlled clinical trial at field site, Howard University Medical Center in Washington, DC, involving 138 older African American men and women (55 years of age and older) with documented atherosclerotic CVD who will be randomized to supplementation with either the traditional CAM herbal preparation (MAK 4+5), conventional vitamin cocktail (E+C) or placebo for 12 months. Clinical and mechanistic outcomes include carotid artery atherosclerosis (IMT), endothelial dysfunction (brachial artery reactivity), oxidized LDL, traditional CVD risk factors (BP, lipids, diet, exercise, smoking, weight) and quality of life. Participants will continue usual care. The results of this clinical study will provide much needed understanding of the basic and clinical effects of a traditional herbal antioxidant preparation on pathophysiological mechanisms of atherosclerotic CVD in this high risk group. This will facilitate translation of research findings on CAM into clinical practice for prevention of disease in this underserved and understudied population of high risk older African Americans.

ELIGIBILITY:
Inclusion Criteria:

* African American (self-identified)
* Atherosclerotic coronary heart disease (CHD)defined by documented clinical history of myocardial infarction, coronary revascularization procedure (CABG, PTCA), or coronary angiography demonstrating at least one coronary artery with >50% stenosis
* High risk for CVD, defined as >=2 on Framingham/ATP III risk factor scale
* Informed consent
* Written permission of participant's referring physician

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 1999-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Schneider, Principal Investigator — Center for Health and Aging Studies
Locations (2):
- United States (2):
  - Howard University Medical Center, Washington D.C., District of Columbia
  - Maharishi University of Management, Fairfield, Iowa